CLINICAL TRIAL: NCT00412334
Title: Antiviral Effect of 4 Regimens of PEGASYS Plus Copegus in Patients With Genotype 1 Chronic Hepatitis C Non-responder to Previous Peginterferon Alfa-2a Plus Ribavirin Therapy
Brief Title: SYREN Study: A Study of PEGASYS (Peginterferon Alfa-2a (40KD)) Plus Copegus (Ribavirin) in Non-Responder Patients With Chronic Hepatitis C (CHC) Genotype 1.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20399
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2a

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Copegus; Drug: peginterferon alfa-2a [Pegasys]
- 2 (Experimental)
  Interventions: Drug: Copegus; Drug: peginterferon alfa-2a [Pegasys]
- 3 (Experimental)
  Interventions: Drug: Copegus; Drug: peginterferon alfa-2a [Pegasys]
- 4 (Experimental)
  Interventions: Drug: Copegus; Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: Copegus — 1200-1600mg/day po
  Arms: 3; 4
Drug: Copegus — 1000-1200mg/day po
  Arms: 1; 2
Drug: peginterferon alfa-2a [Pegasys] — 360 micrograms sc weekly
  Arms: 1; 3
Drug: peginterferon alfa-2a [Pegasys] — 180 micrograms sc twice weekly
  Arms: 2; 4

SUMMARY:
This study will evaluate the efficacy and safety of 4 regimens of PEGASYS plus Copegus, in patients with chronic hepatitis C (CHC) genotype 1 who have failed to respond to previous treatment with standard doses of PEGASYS plus ribavirin. Patients will be randomized to one of 4 groups, to receive a)PEGASYS 360 micrograms/week plus Copegus 1000-1200mg/day, b)PEGASYS 180 micrograms twice weekly plus Copegus 1000-1200mg/day, c)PEGASYS 360micrograms/week plus Copegus 1200-1600mg/day, or d)PEGASYS 180 micrograms twice weekly plus Copegus 1200-1600mg/day. Following 48 weeks treatment, there will be a 24 week period of treatment-free follow-up. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age, with CHC genotype 1;
* patients who have failed to respond to previous treatment with PEGASYS plus ribavirin for >=12 weeks;
* patients who have discontinued PEGASYS/ribavirin >=4 weeks prior to enrollment;
* compensated liver disease.

Exclusion Criteria:

* other forms of liver disease;
* infection with HIV, HAV, HBV;
* hepatocellular cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2007-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Sustained viral response | Week 72

SECONDARY OUTCOMES:
Percentage of patients with >=2log drop of HCV-RNA | Week 4, 12, 24.
Percentage of patients with non-detectable HCV-RNA | Week 48
Relapse rate | Throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- France (19):
  - Angers
  - Bobigny
  - Châteauroux
  - Créteil
  - Grenoble
  - Hyères
  - Lille
  - Limoges
  - Marseille
  - Metz
  - Montpellier
  - Nice
  - Paris
  - Pessac
  - Poitiers
  - Strasbourg
  - Toulouse
  - Vandœuvre-lès-Nancy
  - Villejuif

REFERENCES:
- [Derived] Chevaliez S, Hezode C, Soulier A, Costes B, Bouvier-Alias M, Rouanet S, Foucher J, Bronowicki JP, Tran A, Rosa I, Mathurin P, Alric L, Leroy V, Couzigou P, Mallat A, Charaf-Eddine M, Babany G, Pawlotsky JM. High-dose pegylated interferon-alpha and ribavirin in nonresponder hepatitis C patients and relationship with IL-28B genotype (SYREN trial). Gastroenterology. 2011 Jul;141(1):119-27. doi: 10.1053/j.gastro.2011.03.039. Epub 2011 Mar 24. PMID 21439960